CLINICAL TRIAL: NCT01157221
Title: Determining Shoulder Kinematics in the Prediction of Progress of Frozen Shoulder Syndrome: a Prediction Method, Validation of the Method, and Clinical Application
Brief Title: Prediction Frozen Shoulder Validation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, School of Physical Therapy, National Taiwan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 200612088R
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-06

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intervention group (Experimental): intervention group: end-range mobilization/scapular mobilization treatment approach group
  Interventions: Other: EMSMTA
- control (Active Comparator)
  Interventions: Other: a standardized physical therapy program
- control-criteria group (Sham Comparator)
  Interventions: Other: a standardized physical therapy program

INTERVENTIONS:
Other: a standardized physical therapy program — passive mobilization, stretching techniques, physical modalities (i.e., ultrasound, shortwave diathermy, and/or electrotherapy), and active exercises
  Arms: control; control-criteria group
Other: EMSMTA — end-range mobilization/scapular mobilization treatment approach
  Arms: intervention group

SUMMARY:
Background: Few studies have examined the predictors of the clinical course of subjects with frozen shoulder syndrome or explained the persistence of symptoms after appropriate therapy. Altered shoulder kinematics may predispose subjects to subacromial impingement, rotator cuff tendonitis, altered shoulder joint forces, and possible degenerative changes. Subsequently, a more difficult and chronic course of frozen shoulder syndrome may develop.

Objective: The purposes of this study are: (1) to develop a prediction method for determining altered shoulder kinematics and associated muscular activities which are associated with the chronicity of frozen shoulder dysfunction, and (2) to validate this prediction method and analyze the impact of the method on clinical behavior.

Design: For the first year, a prospective study will be conducted to develop a prediction method that will identify impaired shoulder kinematics associated with the degree of symptom-related functional disability in patients with frozen shoulder syndrome. For the second and third years, validation of the proposed prediction method will determine whether altered shoulder kinematics and associated muscular activities subject to intervention meet the prediction criteria and demonstrate improvement in their follow-up, which will be shown to improve decision making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 50% loss of passive movement of the shoulder joint relative to the nonaffected side, in 1 or more of 3 movement directions (i.e., forward flexion, abduction in the frontal plane, or external rotation in 0° of abduction);
* 13-15 and duration of complaints of at least 3 months.

Exclusion Criteria:

* a history of stroke with residual upper-extremity involvement,
* diabetes mellitus,
* rheumatoid arthritis,
* rotator cuff tear,
* surgical stabilization of the shoulder,
* osteoporosis, or
* malignancies in the shoulder region.
* subjects who had pain or disorders of the cervical spine, elbow, wrist, or hand, or who had pain radiating from the shoulder to the arm, were also excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Range of motion | pre 4 weeks 8 weeks
Disability assessment | pre 4 weeks 8 weeks
Shoulder complex kinematics | pre 4 weeks 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jiu-jenq Lin, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan